CLINICAL TRIAL: NCT03498105
Title: Utility of the Cardiac Electrical Biomarker in Patients With Ischaemic Heart Disease
Brief Title: Utility of the Cardiac Electrical BiomarkerDisease
Acronym: VECTRA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Joanne Turner (Other Government)
Responsible Party: Sponsor-Investigator, Joanne Turner, Academic Research Coordinator, Milton Keynes University Hospital NHS Foundation Trust
Organization: Milton Keynes University Hospital NHS Foundation Trust (Other Government)
Other Study IDs: 16-MK-008
Record Dates: First submitted 2017-09-08; First posted 2018-04-13 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Acute Chest Syndrome
Keywords: Acute Chest Syndrome
MeSH Terms: conditions — Acute Chest Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Emergency Department (ED): 450-500 participants who will;
  1. self present to the Emergency Department (ED) will chest pain
  2. be brought in by ambulance to ED with acute chest pain
  3. be referred from Primary care or Urgent care centre with cardiac sounding chest pain
- Community Cardiology Service (CCS): This study group will consist of between 80-100 participants who self present to the Community Cardiology Service (CCS) in Milton Keynes primary care surgery
- Participants with stable angina: This study group will consist of 450-500 participants with stable angina who have been referred for Stress Echocardiography.
- Elective Coronary Angioplasty: This study group will consist of between 50-100 participants who will have been referred for elective coronary angioplasty
- Cardio-toxic Chemotherapy: Consecutive patients being initiated on any of the following medication deemed as cardio toxic and requiring cardiac function will be approached to be recruited into the study.
- Invasive Coronary Angiography: The dynamics and performance characteristics of the CEB during acute coronary occlusion in patients undergoing invasive coronary angiography.

SUMMARY:
This project is aiming to identify the diagnostic utility CEB (Cardiac Electrical Biomarker) in patients who are undergoing cardiac investigations.

DETAILED DESCRIPTION:
This project is aiming to identify the diagnostic utility of an ECG derived measurement by a Medical device (Vectraplex by VectraCor ltd) in patients who are undergoing cardiac investigations. This technology is based on the principle of vector ECG and an analysing system that computes a composite score termed a Cardiac Electrical Biomarker (CEB TM).

CEB has been validated in the detection of STEMI with high sensitivity and specificity in the detection ECG changes characteristic to STEMI. The CEB may be a more accurate way of identifying heart injury and causes of chest pain compared to standard tests, which could lead to faster diagnosis and treatment of these patients.

The diagnostic utility of the CEBTM in the following:

1. Acute chest pain assessment in the A&E department.
2. Acute chest pain assessment in the Primary Care Surgery.
3. Performance of CEB during inducible ischaemia in patients with stable angina
4. Performance of CEB during acute ischaemia in patients undergoing percutaneous coronary intervention (PCI)
5. Performance of CEB in patients undergoing cardio-toxic treatment

ELIGIBILITY:
1. Acute chest pain assessment in the Emergency department

   Inclusion criteria
   * Participant is willing and able to give informed consent for participation in the study
   * Male or Female, aged 18 years or above

   Exclusion criteria

   The participant may not enter the study if ANY of the following apply:
   * Unable or unwilling to give valid consent for participation in the study
   * Participant has been previously recruited to another module of the VECTRA ECG study
   * Participant has history of allergy to ECG electrode
   * Noisy ECG trace in spite of appropriate preparation and elimination of mains artefact and muscle tremor
   * ECG tracing with a wandering baseline
   * Sustained or non-sustained ventricular/atrial arrhythmia (Ventricular tachycardia, supraventricular tachycardia, atrial fibrillation, bigeminy and trigeminy)
   * QRS duration greater than 120 milliseconds
   * Q waves (except positional Q waves checked by deep inspiration)
   * Suspected Septicaemia, pulmonary embolism or aortic dissection
   * Recent history of trauma to thorax
   * Severe renal impairment with eGFR <30 ml/min
2. Acute chest pain assessment in the Primary Care Surgery

   Inclusion criteria
   * Participant is willing and able to give informed consent for participation in the study.
   * Male or Female, aged 18 years or above.
   * Participants who have experienced chest pain more than 6 hours but less than 2 weeks of presentation to the surgery

   Exclusion criteria

   The participant may not enter the study if ANY of the following apply:
   * Unable or unwilling to give valid consent for participation in the study
   * Participant has been previously recruited to another module of the VECTRA ECG study
   * Participant has history of allergy to ECG electrode
   * Participants who have experienced 'Acute chest pain', defined as chest pain occurring less than 6 hours prior to presentation at the surgery
   * Participants whose initial Electrocardiogram reveals features compatible of ST elevation Myocardial Infarction
   * Participants whose initial Electrocardiogram reveals a Left Bundle branch block suspected to be of new onset
   * Noisy ECG trace in spite of appropriate preparation and elimination of mains artefact and muscle tremor
   * ECG tracing with a wandering baseline
   * Sustained or non-sustained ventricular/atrial arrhythmia (Ventricular tachycardia, Supraventricular tachycardia, atrial fibrillation, bigeminy and trigeminy)
   * QRS duration greater than 120 milliseconds
   * Q waves (except positional Q waves checked by deep inspiration)
   * Suspected Septicaemia, pulmonary embolism or aortic dissection
   * Recent history of trauma to thorax
   * Severe renal impairment with eGFR <30ml/min
3. Performance of CEB during inducible ischaemia in patients with stable angina

   Inclusion criteria
   * Participant is willing and able to give informed consent for participation in the study.
   * Male or Female, aged 18 years or above.

   Exclusion criteria

   The participant may not enter the study if ANY of the following apply:
   * Unable or unwilling to give valid consent for participation in the study
   * Participant has been previously recruited to another module of the VECTRA ECG study
   * Lack of adequate ultrasound acoustic window
   * Contraindications to undergoing stress test using dobutamine
   * Participant has history of allergy to ECG electrode
   * Noisy ECG trace in spite of appropriate preparation and elimination of mains artefact and muscle tremor
   * ECG tracing with a wandering baseline
   * Sustained or non-sustained ventricular/atrial arrhythmia (Ventricular tachycardia, supraventricular tachycardia, atrial fibrillation, bigeminy and trigeminy)
   * QRS duration greater than 120milliseconds
   * Q waves (except positional Q waves checked by deep inspiration)
   * Suspected Septicaemia, pulmonary embolism or aortic dissection
   * Recent history of trauma to thorax
   * Severe renal impairment with eGFR <30 ml/min
4. Performance of CEB during acute ischaemia in patients undergoing percutaneous coronary intervention (PCI)

   Inclusion criteria
   * Participant is willing and able to give informed consent for participation in the study
   * Male or Female, aged 18 years or above
   * Participant diagnosed with stable CAD or stable ACS (unstable angina or NSTEMI with no pulmonary oedema or cardiogenic shock at the time of recruitment)
   * Participant with Single vessel coronary artery disease or multi- vessel disease for target vessel PCI

   Exclusion criteria

   The participant may not enter the study if ANY of the following apply:
   * Unable or unwilling to give valid consent for participation in the study
   * Participant has been previously recruited to another module of the VECTRA ECG study
   * Participant has history of allergy to ECG electrode
   * Participants known to have multi-vessel coronary artery disease with one or more Chronic Total Occlusive lesions
   * Severe Left main coronary artery stenosis
   * Noisy ECG trace in spite of appropriate preparation and elimination of mains artefact and muscle tremor
   * ECG tracing with a wandering baseline
   * Sustained or non-sustained ventricular/atrial arrhythmia (Ventricular tachycardia, supraventricular tachycardia, atrial fibrillation, bigeminy and trigeminy)
   * QRS duration greater than 120 milliseconds
   * Q waves (except positional Q waves checked by deep inspiration)
   * Suspected Septicaemia, pulmonary embolism or aortic dissection
   * Recent history of trauma to thorax
   * Severe renal impairment with eGFR <30 ml/min
5. Performance of CEB in patients undergoing cardio-toxic treatment (type 1 and type 2 cytostatic based treatments of haemo-oncological patients

Inclusion criteria

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Participants who have been given a diagnosis of cancer and are being commenced on a chemotherapeutic drug deemed to be cardio-toxic

Exclusion criteria

The participant may not enter the study if ANY of the following apply:

* Unable or unwilling to give valid consent for participation in the study
* Participant has been previously recruited to another module of the VECTRA ECG study
* Participant has history of allergy to ECG electrode
* Participants previously diagnosed with Cardiomyopathy or Heart failure
* Lack of adequate ultrasound acoustic window
* Noisy ECG trace in spite of appropriate preparation and elimination of mains artefact and muscle tremor
* ECG tracing with a wandering baseline
* Sustained or non-sustained ventricular/atrial arrhythmia (Ventricular tachycardia, supraventricular tachycardia, atrial fibrillation, bigeminy and trigeminy)
* QRS duration greater than 120milliseconds
* Q waves (except positional Q waves checked by deep inspiration)
* Suspected Septicaemia, pulmonary embolism or aortic dissection
* Recent history of trauma to thorax
* Severe renal impairment with eGFR <30ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing investigations for Ischaemic heart disease and cardio-toxic effects of chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2017-05-22 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of CEB in detecting myocardial injury | Day 1
  Metrics: sensitivity, specificity, PPV, NPV

SECONDARY OUTCOMES:
Correlation between CEB and cardiovascular mortality | 30 days and 12 months
  Cardiovascular death
Correlation between CEB and non-fatal myocardial infarction | 30 days and 12 months
  Non-fatal myocardial infarction
Correlation between CEB and readmission with progressive angina | 30 days and 12 months
  Readmission with angina after index admission
Relationship between CEB and need for revascularisation | 30 days and 12 months
  Revascularisation (surgery or Percutaneous Coronary Intervention) from index admission

CONTACTS AND LOCATIONS:
Overall Officials: Attila kardos, Principal Investigator — Milton Keynes University Hospital NHS Foundation Trust
Locations (1):
- Milton Keynes University Hospital NHS Foundation Trust, Milton Keynes, Bucks, United Kingdom

IPD SHARING:
Plan to Share IPD: No